CLINICAL TRIAL: NCT02575313
Title: The Effects of Whole Food Intervention on Mucositis in Patients Being Treated for Head and Neck Cancer With Radiation With or Without Chemotherapy
Brief Title: The Effects of Whole Food Intervention on Mucositis in Patients Treated for Head and Neck Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of participant recruitment.
Sponsor: Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-173B
Record Dates: First submitted 2015-09-25; First posted 2015-10-14 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Mucositis
Keywords: L-Glutamine; chemotherapy; radiotherapy; therapeutic toxicity
MeSH Terms: conditions — Mucositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Whole Food Intervention Treated (Experimental): Group of participants given the experimental WFI along with standard cancer treatment.
  Interventions: Dietary Supplement: Whole Food Intervention

INTERVENTIONS:
Dietary Supplement: Whole Food Intervention — A combination of honey, glutamine, probiotics, and butter was administered to participants undergoing cancer.

SUMMARY:
This is a study to see if a Whole Food Intervention (WFI) consisting of yogurt, butter, honey, vanilla, and glutamine will lower the frequency or severity of mucositis in head and neck cancer patients undergoing standard treatment.

DETAILED DESCRIPTION:
The proposal is a one center, open label, randomized pilot study to evaluate the safety, tolerability and compliance of a Whole Food Intervention with Standard of Care for patients with head & neck cancer. The primary objectives are:

1. To determine whether patients will use a Whole Food Intervention 4-6 times daily, and
2. To determine whether the Whole Food Intervention will reduce the incidence of grade 2 or greater mucositis from 75% historically seen to 25% .
3. To determine whether Whole Food Intervention will reduce the incidence of treatment breaks from >19% to < 10% (see section 9 for comments)

This Whole Food Intervention will be taken by mouth before the start of radiation therapy, with or without chemotherapy and for the entire treatment therapy.

Mucositis-related pain and reduction of oral intake will be quantified by using validated assessment tools. Weight loss or gain, diarrhea, constipation or no change in bowel function and the use of conventional medication for radiation-induced mucositis will be recorded. Chart review and patient questionnaires will be used to establish whether a treatment break or dose reduction for radiation of chemotherapy was required due to radiation mucositis-related symptoms. Complete Chemistry Profile and Complete Blood Count will be extracted from the patients' medical oncologist's or radiation oncologist's records. The patient will continue to use standard mucositis therapies if desired as prescribed by the treating oncology physician.

The Whole Food Intervention consists of yogurt, butter, honey, vanilla, and glutamine with 3 portioning cups, equal to approximately 12 ounces, taken daily before starting radiation therapy. A questionnaire will be used to record symptoms and doses taken. The patient will continue to use standard mucositis therapies as prescribed by the treating oncology physician.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed diagnosis of head & neck carcinoma
* Scheduled to undergo continuous daily course of radiation therapy with or without chemotherapy
* No other serious concurrent medical illness as determined by the Principle Investigator
* Absolute neutrophil count ≥ 500/mm3
* Platelet count ≥ 50,000/mm3
* No history of insulin-dependent diabetes mellitus
* No prior hypersensitivity reaction to compound components

Exclusion Criteria:

* Dislike of the available forms of the WFI
* Allergy or food intolerance relevant to the ingredients
* Lack of access to refrigerated storage for the WFI
* Inability or unwillingness to participate twice a week
* Inability to swallow
* Undergoing treatment for HIV with HIV medications
* Ongoing alcohol and/or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Measurement of Tolerability | Eight (8) weeks
  Estimated portion consumption on a daily basis was obtained to determine if the WFI could be tolerated by participants.

SECONDARY OUTCOMES:
Mucositis Grading | Eight (8) weeks
  Mucositis grade was calculated using established criteria.
Treatment Break Measurement | Eight (8) weeks
  To determine whether Whole Food Intervention will reduce the incidence of treatment breaks from ≥19% to ≤10%.

CONTACTS AND LOCATIONS:
Overall Officials: Miles H Hassell, MD, Principal Investigator — Providence Health & Services
Locations (2):
- United States (2):
  - The Oregon Clinic, Providence Portland Cancer Center, Portland, Oregon
  - Integrative Medicine Program, Providence St. Vincent Medical Center, Portland, Oregon